CLINICAL TRIAL: NCT05657574
Title: A Randomized, Double-blind, Multi-center, Therapeutic Confirmatory, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-391 and CKD-331 in Patients With Primary Hypercholesterolemia
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of CKD-391 and CKD-331 in Patients With Primary Hypercholesterolemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A52_08HCL2217
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CKD-391 (Experimental): D377 + CKD-331 + placebo (for D086)
  Interventions: Drug: D377; Drug: CKD-331; Drug: Placebo (for D086)
- CKD-331 (Active Comparator): CKD-331 + placebo (for D377) + placebo (for D086)
  Interventions: Drug: CKD-331; Drug: Placebo (for D377); Drug: Placebo (for D086)
- D377 (Active Comparator): D377 + placebo (for CKD-331) + placebo (for D086)
  Interventions: Drug: D377; Drug: Placebo (for CKD-331); Drug: Placebo (for D086)
- D086 (Active Comparator): D086 + placebo (for D377) + placebo (for CKD-331)
  Interventions: Drug: D086; Drug: Placebo (for D377); Drug: Placebo (for CKD-331)

INTERVENTIONS:
Drug: D377 — oral, once daily, 8 weeks
  Arms: CKD-391; D377
Drug: CKD-331 — oral, once daily, 8 weeks
  Arms: CKD-331; CKD-391
Drug: D086 — oral, once daily, 8 weeks
  Arms: D086
Drug: Placebo (for D377) — oral, once daily, 8 weeks
  Arms: CKD-331; D086
Drug: Placebo (for CKD-331) — oral, once daily, 8 weeks
  Arms: D086; D377
Drug: Placebo (for D086) — oral, once daily, 8 weeks
  Arms: CKD-331; CKD-391; D377

SUMMARY:
This is a randomized, double-blind, multi-center, therapeutic confirmatory, phase 3 trial to evaluate the efficacy and safety of CKD-391 and CKD-331 in patients with primary hypercholesterolemia

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1:1:1 ratio to the following groups: combination therapy of D377 and CKD-331, D377, CKD-331, and D086. The patients are prescribed oral administration of the appropriate IP daily (3 tablets: actual medication and placebo) for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 19 years of age
* Primary hypercholesterolemia
* Patients willing and able to discontinue ongoing lipid-lowering therapy according to the opinion of the investigator

Exclusion Criteria:

* Secondary hypercholesterolemia
* Conditions / situations such as:

  1. Presence of any clinically significant uncontrolled endocrine/metabolic disease known to influence lipids levels
  2. Severe renal impairment or active liver disease
* History of hypersensitivity or allergies to investigational drugs or drug of similar chemical classes.
* History of drug abuse or alcoholism within 24 weeks before screening
* Any surgical or medical condition which might significantly affect the absorption, distribution, metabolism, or excretion of investigational drugs
* Patients who have been taken with other investigational drugs within 8 weeks before screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change | Baseline, Week 8
  from Baseline at Week 8 of Low Density Lipoprotein Cholesterol (LDL-C)

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No